CLINICAL TRIAL: NCT05304455
Title: Apixaban for Prevention of Portal Vein Thrombosis in Liver Cirrhotic Patients After Laparoscopic Splenectomy and Azygoportal Disconnection for Portal Hypertension
Brief Title: Apixaban Prevents Portal Vein Thrombosis After Laparoscopic Splenectomy and Azygoportal Disconnection
Acronym: ESAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Guo-Qing Jiang, Clinical Professor, Northern Jiangsu People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: YZUC-009
Record Dates: First submitted 2022-03-19; First posted 2022-03-31 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Cirrhosis; Splenectomy; Venous Thrombosis; Hypertension, Portal
Keywords: Cirrhosis; Venous thrombosis; Portal Hypertension; Apixaban; Splenectomy; Laparoscopy
MeSH Terms: conditions — Fibrosis; Venous Thrombosis; Hypertension, Portal | interventions — apixaban; Dipyridamole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apixaban group (Experimental): From postoperative day 3, Patients will receive oral Dipyridamole 25mg tid for three months along with subcutaneous Low Molecular Weight Heparin injection for first five days and 2.5 mg oral Apixaban tablets (Bristol-Myers Squibb, Cruiserath, USA) twice daily for 6 months.
  Interventions: Drug: Apixaban 2.5 MG; Drug: Dipyridamole 25Mg Tab; Drug: subcutaneous Low Molecular Weight Heparin

INTERVENTIONS:
Drug: Apixaban 2.5 MG — From postoperative day 3, Patients will receive oral dipyridamole 25mg tid for three months along with subcutaneous Low Molecular Weight Heparin injection for first five days and 2.5 mg oral Apixaban tablets (Bristol-Myers Squibb, Cruiserath, USA) twice daily for 6 months.The Doppler Ultra Sonography screening will be done to assess the occurrence of portal vein thrombus.
  Other Names: ELIQUIS
Drug: Dipyridamole 25Mg Tab — From postoperative day 3, Patients will receive oral dipyridamole 25mg tid for three months along with subcutaneous Low Molecular Weight Heparin injection for first five days and 2.5 mg oral Apixaban tablets (Bristol-Myers Squibb, Cruiserath, USA) twice daily for 6 months.The Doppler Ultra Sonography screening will be done to assess the occurrence of portal vein thrombus.
  Other Names: Persantine
Drug: subcutaneous Low Molecular Weight Heparin — From postoperative day 3, Patients will receive oral dipyridamole 25mg tid for three months along with subcutaneous Low Molecular Weight Heparin injection for first five days and 2.5 mg oral Apixaban tablets (Bristol-Myers Squibb, Cruiserath, USA) twice daily for 6 months.The Doppler Ultra Sonography screening will be done to assess the occurrence of portal vein thrombus.
  Other Names: LMWHs

SUMMARY:
The purpose of this study is to determine whether Apixaban is effective and safe in Prevention of Portal Vein Thrombosis in Liver Cirrhotic Patients after Laparoscopic Splenectomy and Azygoportal Disconnection

DETAILED DESCRIPTION:
After successful screening the cases of cirrhosis of liver irrespective of the etiology who have no portal vein thrombosis will be enrolled. From postoperative day three, patients in apixaban group will receive oral Apixaban 2.5mg bid for six months, and be along with five days of subcutaneous injection of Low Molecular Weight Heparin and three months of oral Dipyridamole. The Doppler screening for the occurrence of portal vein thrombus (PVT) or spleno-mesenteric thrombosis will be done for all patients at baseline, on postoperative months (POD) 7, at postoperative months (POM) 1, 3, and 6. All groups will receive the therapy for six months irrespective of the Doppler findings in relation to portal vein thrombus occurrence. Then six months monitoring will be done as per the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical, radiological or histologic diagnosis of cirrhosis of any etiology
2. Splenomegaly with secondary hypersplenism
3. Bleeding portal hypertension
4. No evidence of PVT or spleno-mesenteric thrombosis by ultrasound evaluation and angio-CT
5. Informed consent to participate in the study

Exclusion Criteria:

1. Hepatocellular carcinoma or any other malignancy,
2. Hypercoagulable state other than the liver disease related
3. DRUGS- oral contraceptives, anticoagulation or anti-platelet drugs.
4. Child - Pugh C
5. Recent peptic ulcer disease
6. History of Hemorrhagic stroke
7. Pregnancy.
8. Uncontrolled Hypertension
9. Human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with Main and Intrahepatic Branches of Portal Vein Thrombosis | 6 months
  Proportion of participants with Main and intrahepatic branches of portal vein thrombosis by ultrasound evaluation

SECONDARY OUTCOMES:
Proportion of participants with Splenic vein thrombosis | 6 months
  Proportion of participants withSplenic vein thrombosis by ultrasound evaluation
Proportion of participants with Mesenteric vein thrombosis | 6 months
  Proportion of participants with Mesenteric vein thrombosis by ultrasound evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Ping Chen, MD, Study Chair — Clinical Medical College, Yangzhou University
Locations (1):
- Clinical Medical College, Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No